CLINICAL TRIAL: NCT03825289
Title: THREAD: A Phase I Trial of Trametinib and Hydroxychloroquine in Patients With Advanced Pancreatic Cancer
Brief Title: Trametinib and Hydroxychloroquine in Treating Patients With Pancreatic Cancer
Acronym: THREAD
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI116898
Record Dates: First submitted 2019-01-30; First posted 2019-01-31 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Metastatic Pancreatic Carcinoma; Stage II Pancreatic Cancer; Stage IIA Pancreatic Cancer; Stage IIB Pancreatic Cancer; Stage III Pancreatic Cancer; Stage IV Pancreatic Cancer; Unresectable Pancreatic Carcinoma
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Hydroxychloroquine; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (trametinib, hydroxychloroquine) (Experimental): Patients receive trametinib PO QD on days 1-28 and hydroxychloroquine PO QD or BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Hydroxychloroquine; Drug: Trametinib

INTERVENTIONS:
Drug: Hydroxychloroquine — Given PO
Drug: Trametinib — Given PO
  Other Names: GSK1120212; JTP-74057; MEK Inhibitor GSK1120212; Mekinist

SUMMARY:
This phase I trial studies the sides effects and best dose of hydroxychloroquine when given together with trametinib in treating patients with pancreatic cancer that has spread to nearby tissue, lymph nodes or other places in the body and cannot be removed by surgery. Trametinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as hydroxychloroquine, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving trametinib together with hydroxychloroquine may work better in treating patients with pancreatic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the recommended phase II dose of hydroxychloroquine in combination with trametinib as assessed by the occurrence of dose-limiting toxicities (DLTs).

ELIGIBILITY:
Inclusion Criteria:

* Subject with histologically confirmed metastatic or locally advanced, unresectable pancreatic carcinoma
* Subject is willing to provide a baseline biopsy.
* EXPANSION COHORT ONLY: Subject must have progressed during or after two standard of care lines of treatment or refused standard of care options.
* Subject must have computed tomography (CT) measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria
* Subject must be able and willing to undergo disease assessment while on study and afterwards, if removed for reason other than progression
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L
* Platelet count >= 100 x 10^9/L
* Hemoglobin >= 9 g/dL
* Total bilirubin level =< 1.5 x the upper limit of normal (ULN) range
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels =< 3 x ULN. Patients with liver metastases will be allowed to enroll with AST and ALT levels =< 5 x ULN
* Estimated creatinine clearance >= 30 mL/min according to the Cockcroft-Gault formula (or local institutional standard method)
* Negative serum or urine pregnancy test at screening for women of childbearing potential
* Highly effective contraception for both male and female subjects throughout the study and for at least 4 months after last study treatment administration
* Recovery to baseline or =< grade 1 Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0 from toxicities related to any prior treatments, unless adverse event (AE)(s) are clinically nonsignificant and/or stable on supportive therapy
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines

Exclusion Criteria:

* Subject who have received systemic antineoplastic therapy (including unconjugated therapeutic antibodies and toxin immunoconjugates) or any investigational therapy within 2 weeks or within 5 half-lives of the investigational therapy prior to starting study treatment, whichever is shorter.
* Subject who have received radiotherapy within 2 weeks prior to the first dose of study treatment. Localized radiation therapy for the treatment of symptomatic bone metastasis is allowed during that timeframe
* Subjects who have undergone major surgery =< 3 weeks prior to starting study drug or who have not recovered from side effects of such procedure
* Patients with multiple primary malignancies may be enrolled if non-pancreatic ductal adenocarcinoma (PDAC) tumor(s) does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen as determined by treating investigator and do not require active treatment
* Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 4 weeks before first dose of study treatment. Eligible subjects must be neurologically asymptomatic and without corticosteroid treatment at the time of first dose of study treatment
* History or current evidence of retinal vein occlusion (RVO) or current risk factors for RVO (e.g. uncontrolled glaucoma or ocular hypertension, history of hyperviscosity or hypercoagulability syndromes)
* History of active major bleeding.
* Patients whom thromboembolic prophylaxis is medically contraindicated per the treating investigator's assessment.
* Current evidence of uncontrolled, significant intercurrent illness including, but not limited to, the following conditions:

  * Cardiovascular disorders:

    * Congestive heart failure New York Heart Association class 3 or 4, unstable angina pectoris, serious cardiac arrhythmias.
    * Stroke (including transient ischemic attack [TIA]), myocardial infarction (MI), or other ischemic event, or thromboembolic event (eg, deep venous thrombosis, pulmonary embolism) within 3 months before first dose. The presence of an asymptomatic portal vein thrombosis will not preclude study participation.
  * History of glucose-6-phosphate dehydrogenase (G6PD) deficiency
  * History of seizures
  * Patients who are planning on embarking on a new strenuous exercise regimen after first dose of study treatment. Muscular activities, such as strenuous exercise, that can result in significant increases in plasma creatine kinase (CK) levels should be avoided while on study treatment
  * Patients who have neuromuscular disorders that are associated with elevated CK (e.g., inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy)
  * Impairment of gastrointestinal function or gastrointestinal disease (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection that under the judgment of the principal investigator [PI] may impair absorption of study drugs)
  * Any other condition that would, in the Investigator?s judgment, contraindicate the patient?s participation in the clinical study due to safety concerns or compliance with clinical study procedures, e.g., infection/inflammation, intestinal obstruction, unable to swallow medication.(patients may not receive drug through a feeding tube), social/ psychological issues, etc
* Screening corrected QT interval by Fridericia (QTcF) > 500 msec
* Known human immunodeficiency virus (HIV), unless patient is on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* Known chronic hepatitis B virus, unless hepatitis B virus (HBV) viral load is undetectable
* Known history of hepatitis C virus (HCV) infection, unless treated and cured; for patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Medical, psychiatric, cognitive or other conditions that may compromise the patient's ability to understand the patient information, give informed consent, comply with the study protocol or complete the study
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test
* Sexually active males who are not willing to use a condom during intercourse while taking the drug and for 4 months after stopping treatment. A condom is also required to be used by vasectomized men in order to prevent delivery of the drug via seminal fluid
* Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (National Cancer institute [NCI] CTCAE v5.0 grade >= 3)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-01-18 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Rate of dose-limiting toxicities during the DLT assessment window. | At 28 days
  To determine the recommended phase II dose (RP2D) hydroxychloroquine in combination with trametinib.

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) for the duration of study treatment | 30 days after last dose
  To assess the safety of the combination of trametinib and hydroxychloroquine
Response Rate | 5 years
  To assess the efficacy of the combination of trametinib and hydroxychloroquine

CONTACTS AND LOCATIONS:
Overall Officials: Conan Kinsey, MD, Principal Investigator — Huntsman Cancer Institute/ University of Utah
Locations (2):
- United States (2):
  - University of California, San Francisco, San Francisco, California
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No